CLINICAL TRIAL: NCT05023655
Title: A Phase II Study of Tazemetostat in Solid Tumors Harboring an ARID1A Mutation
Brief Title: Phase II Study of Tazemetostat in Solid Tumors Harboring an ARID1A Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPZ-IST-001
Record Dates: First submitted 2021-08-12; First posted 2021-08-26 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; ARID1A Gene Mutation
Keywords: ARID1A mutation; solid tumors; tazemetostat
MeSH Terms: interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tazemetostat (Experimental): tazemetostat 800 mg po twice daily in continuous 28- day cycles
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — 800mg po twice daily
  Other Names: tazverik

SUMMARY:
The FDA approved targeted agent tazemetostat inhibits EZH2 and induces durable tumor responses in patients with B-cell non-Hodgkin's lymphoma and epithelioid sarcomas. Responses have also been demonstrated in INI1 and SMARCA4 negative solid tumors patients. Since EZH2 plays a critical role in driving the biology of ARID1A mutated malignancies, we hypothesize that inhibition of EZH2 with tazemetostat will lead to significant clinical benefit in ARID1A mutated malignancies.

DETAILED DESCRIPTION:
AT rich interacting domain containing protein 1A (ARID1A) is a tumor suppressor gene frequently mutated in solid tumor malignancies, often loss of function mutations (frameshift or non-sense). ARID1A encodes a large nuclear protein BAF250a, a vital component of the Switch/Sucrose Non-Fermentable (SWI/SNF) chromatin remodeling complex, which participates in several nuclear activities including transcription, DNA synthesis and DNA damage repair. ARID1A alterations are particularly prevalent in ovarian clear cell carcinoma (46-50%), ovarian and uterine endometrioid carcinomas (24-44%), and cholangiocarcinoma (27%); reported in up to 27% of gastric carcinoma, esophageal adenocarcinoma, Waldenstrom macroglobulinemia, pediatric Burkitt lymphoma, hepatocellular carcinoma, urothelial carcinoma, 12% of colorectal carcinoma (CRC) , 15% of invasive ductal carcinoma of breast, and 7.5% of NSCLC, as a sample representation reported in the COSMIC database.

ARID1A plays a key role in regulating cell cycle and DNA damage repair, through its critical role in chromatin regulation. Loss of function of ARID1A leads to dysregulation of many gene pathways, supporting its role as a tumor suppressor gene. Loss of ARID1A mediates fulvestrant resistance, demonstrated in multiple elegant studies involving ER+ breast cancer lines, related to therapeutic pressure and selection [1]. Sporadic deletion of ARID1A in mice leads to de novo invasive colon adenocarcinoma. Loss of ARID1A leads to deregulation of the MEK/ERK pathway, critical in kras mutated CRC. ARID1A loss is associated with microsatellite instability in ovarian and endometrial endometrioid adenocarcinomas and gastric cancer. Preclinical data demonstrates enhanced clinical activity of check point inhibitors in ARID1A mutated tumors.

EZH2, enhancer of zeste homologue 2, the enzymatically active core of PRC2 (polycomb repression complex 2/3) plays a key role in tumorigenesis. Over-expression in tumor cells leads to histone hypermethylation, tumor proliferation, cell cycle dysregulation, metastases and angiogenesis.

Tazemetostat is an FDA approved selective small molecule inhibitor of the histone lysine methyltransferase enhancer of zeste homolog 2 (EZH2). Posttranslational modifications of core histone proteins of chromatin play an important role in controlling the fidelity of gene transcription patterns in cells. Paramount among these transcription-controlling modifications is methylation events at lysine and arginine residues, catalyzed by histone methyltransferases (HMTs). Genetic alterations in a number of HMTs have been identified in human cancers where they are purported to play a causal role in malignancies. Tazemetostat has been shown to produce durable tumor responses in patients with B-cell non-Hodgkin's lymphoma and epithelioid sarcomas. Responses have also been demonstrated in INI1 and SMARCA4 negative solid tumors patients.

Hypothesis: EZH2 plays a critical role in driving the biology of ARID1A mutated malignancies. Inhibition of EZH2 with tazemetostat will lead to significant clinical benefit in ARID1A mutated malignancies.

Cell homeostasis requires a balance in ARID1A and EZH2 through chromatin mediated gene expression. Loss of ARID1A expression leads to imbalance, with enhanced EZH2 activity in malignancies. Targeted EZH2 inhibition in ARID1A mutated tumors leads to synthetic lethality in several malignancies, with upregulation of PI3K interacting protein 1 gene (PI3K1P1) and associated growth suppression. EZH2 plays a key role in ovarian carcinoma. Benjamin Bitler et al [2] demonstrated PIK3IP1 as a direct target of ARID1A and EZH2, upregulated by EZH2 inhibition and contributing to synthetic lethality by inhibiting PI3K-AKT signaling. EZH2 inhibition caused in vivo regression of ARID1A-mutated ovarian tumors. A recent published study suggests the synthetic lethality of targeting EZH2 in ARID1A mutated gastric cancer. Leo Yamada et al [3] demonstrated selective sensitivity of EZH2 inhibitors against ARID1A-deficient GC supporting the potential efficacy of targeted therapy using EZH2 inhibitors in this patient population. Targeting EZH2 has also demonstrated potential synthetical lethality in kras mutated CRC in ARID1A mutated tumors [4].

The Prisma Health Cancer Institute reviewed molecular profiling of current patients and identified 124 cancer patients with an ARID1A mutation in a spectrum of malignancies including breast, non-small cell lung cancer, pancreas, uterine, ovarian, cholangiocarcinoma, hepatocellular, and multiple rare solid tumors. A high frequency of concurrent PTEN and PI3K pathways mutations along with ARID1A mutations was also seen, suggesting a potentially significant role of EZH2.

There are no clinical trials addressing therapy in ARID1A mutated malignancies. A current clinical trial, NCT03348631, is evaluating tazemetostat in patients with recurrent ovarian, peritoneal, and endometrial cancer, not selected by ARID1A mutation status [5].

These data support the need for further clinical investigation of tazemetostat as monotherapy and in combination with other agents in solid tumors harboring an ARID1A mutation.

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily agreed to provide written informed consent and demonstrated willingness and ability to comply with all aspects of the protocol.
* Histologically and/or cytologically confirmed advanced or metastatic solid tumor harboring ARID1A mutation (except epithelioid sarcoma)
* Progression of disease following approved therapies or for which no standard therapy exists
* For subjects who have experienced any clinically significant toxicity related to a prior anticancer treatment (i.e., chemotherapy, immunotherapy, and/or radiotherapy): at the time the subject provides voluntary written informed consent, all toxicities have either resolved to grade 1 per NCI CTCAE Version 5.0 [11] OR are clinically stable and no longer clinically significant.
* Have measurable disease as defined by RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Males or females are >18 years of age at the time of providing voluntary written informed consent.
* Life expectancy >3 months before enrollment.
* Time between prior anticancer therapy and first dose of tazemetostat as follows:

Cytotoxic chemotherapy - At least 21 days Noncytotoxic chemotherapy (e.g., small molecule inhibitor) - At least 14 days. Nitrosoureas - At least 6 weeks. Monoclonal antibody - At least 28 days. Radiotherapy - At least 14 days. In addition, at least 6 weeks from prior radioisotope therapy; and at least 12 weeks from 50% pelvic or total body irradiation.

* Adequate renal function: Creatinine < 2.0 or calculated creatinine clearance ≥ 35 mL/minute per the Cockcroft and Gault formula
* Adequate bone marrow function:

ANC ≥ 750mm3 without growth factor support (filgrastim or pegfilgrastim) for at least 14 days.

Platelets ≥ 75,000mm3 (≥75 × 109/L) evaluated at least 7 days after platelet transfusion.

Hemoglobin ≥9.0 g/dL and may receive transfusion Adequate liver function: Total bilirubin <1.5 × the upper limit of normal (ULN) (except for unconjugated hyperbilirubinemia of Gilbert's syndrome); Alkaline phosphatase (ALP) (in the absence of bone disease), ALT, and AST <3 × ULN (or <5 × ULN if subject has liver metastases).

Exclusion Criteria:

* Subjects with epithelioid sarcoma are excluded.
* Has a prior history of T-Cell Lymphoblastic Lymphoma, T-Cell Acute Lymphoblastic Leukemia, Myelodysplastic Syndrome, Acute Myeloid Leukemia, or Myeloproliferative Neoplasm.
* Female subjects who are pregnant or breastfeeding.
* Prior exposure to tazemetostat or other inhibitor(s) of EZH2.
* Subjects with uncontrolled CNS metastases requiring steroids.
* Subjects taking medications that are known potent CYP3A4 inducers/inhibitors (including St. John's wort)
* Are unwilling to exclude Seville oranges, grapefruit juice, AND grapefruit from their diet.
* Major surgery within 4 weeks before the first dose of study drug. NOTE: Minor surgery (e.g., minor biopsy of extracranial site, central venous catheter placement, shunt revision) is permitted within 1 week prior to enrollment.
* Are unable to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, vomiting) that might impair the bioavailability of tazemetostat.
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II (Appendix 3), uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac ventricular arrhythmia.
* Have an active infection requiring systemic therapy.
* Known hypersensitivity to any component of tazemetostat.
* Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the subject's participation in this study OR interfere with their ability to receive study treatment or complete the study.
* Subjects who have undergone a solid organ transplant.
* Prior malignancy in the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | through study completion, estimated to be 1 year after the last subject enrolled
  Evidence of anti-tumor activity will be assessed by objective response, as defined by RECIST 1.1. This will be used to summarize ORR (CR+PR), as well as the rates for the individual categories of response, (i.e., CR, PR, SD, and PD).

SECONDARY OUTCOMES:
Disease Control Rate | through study completion, estimated to be 1 year after the last subject enrolled
  DCR defined as the proportion of subjects with best overall response of CR, PR, or SD lasting 3 or more months.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Chung, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health Cancer Institute, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make data available once request is reviewed and approved by the investigators.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: beginning 6 months following publication of study results and ending 24 months post publication
Access Criteria: Data request must be submitted to the principal investigator, reviewed and approved by the study investigators.

REFERENCES:
- [Background] Xu G, Chhangawala S, Cocco E, Razavi P, Cai Y, Otto JE, Ferrando L, Selenica P, Ladewig E, Chan C, Da Cruz Paula A, Witkin M, Cheng Y, Park J, Serna-Tamayo C, Zhao H, Wu F, Sallaku M, Qu X, Zhao A, Collings CK, D'Avino AR, Jhaveri K, Koche R, Levine RL, Reis-Filho JS, Kadoch C, Scaltriti M, Leslie CS, Baselga J, Toska E. ARID1A determines luminal identity and therapeutic response in estrogen-receptor-positive breast cancer. Nat Genet. 2020 Feb;52(2):198-207. doi: 10.1038/s41588-019-0554-0. Epub 2020 Jan 13. PMID 31932695
- [Background] Bitler BG, Aird KM, Garipov A, Li H, Amatangelo M, Kossenkov AV, Schultz DC, Liu Q, Shih IeM, Conejo-Garcia JR, Speicher DW, Zhang R. Synthetic lethality by targeting EZH2 methyltransferase activity in ARID1A-mutated cancers. Nat Med. 2015 Mar;21(3):231-8. doi: 10.1038/nm.3799. Epub 2015 Feb 16. PMID 25686104
- [Background] Yamada L, Saito M, Thar Min AK, Saito K, Ashizawa M, Kase K, Nakajima S, Onozawa H, Okayama H, Endo H, Fujita S, Sakamoto W, Saze Z, Momma T, Mimura K, Ohki S, Kono K. Selective sensitivity of EZH2 inhibitors based on synthetic lethality in ARID1A-deficient gastric cancer. Gastric Cancer. 2021 Jan;24(1):60-71. doi: 10.1007/s10120-020-01094-0. Epub 2020 Jun 6. PMID 32506298
- [Background] Sen M, Wang X, Hamdan FH, Rapp J, Eggert J, Kosinsky RL, Wegwitz F, Kutschat AP, Younesi FS, Gaedcke J, Grade M, Hessmann E, Papantonis A, Strӧbel P, Johnsen SA. ARID1A facilitates KRAS signaling-regulated enhancer activity in an AP1-dependent manner in colorectal cancer cells. Clin Epigenetics. 2019 Jun 19;11(1):92. doi: 10.1186/s13148-019-0690-5. PMID 31217031
- [Background] Campo E, Swerdlow SH, Harris NL, Pileri S, Stein H, Jaffe ES. The 2008 WHO classification of lymphoid neoplasms and beyond: evolving concepts and practical applications. Blood. 2011 May 12;117(19):5019-32. doi: 10.1182/blood-2011-01-293050. Epub 2011 Feb 7. PMID 21300984